CLINICAL TRIAL: NCT00336310
Title: A Double-Blind, Randomized, Parallel, Comparative Study to Evaluate the Efficacy and Safety of an Antidiabetic Agent Repaglinide for the Treatment of Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSRE0001
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2006-06-13 (Estimated); Status verified 2006-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Treatment; Repaglinide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — repaglinide

INTERVENTIONS:
Drug: Repaglinide

SUMMARY:
The purpose of this study is to determine whether a new-brand of repaglinide is effective in the treatment of type 2 diabetes patients.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of a new-brand of repaglinide X® in comparison to Novonorm® for the treatment of type 2 diabetes mellitus patients. Mentally competent patients with age of 30 to 75 years old in Taiwan of either sex with type 2 diabetes mellitus will be included. All eligible subjects will be randomized into treatment groups in 1:1 ratio. The treatment will consist of either X® or Novonorm® tid before meal for 12 weeks of treatment. The primary endpoints include the net change of HbA!c, fasting plasma glucose(FPG)and postprandial plasma glucose(PPG)at the end of 12th week evaluation compared to the baseline visit. Also, safety profiles including adverse event (such as hypoglycemia) incidences, blood pressure, liver, kidney function test will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults of either sex with age 30-75 years old
* Patients have type 2 diabetes mellitus diagnosed after 25 years of age
* Patients have been in poor glycemic control by diet or exercise for at least 1 month or by a stable dose of metformin for at least 3 months before study; poor glycemic control is defined as: Glycosylated hemoglobin A1c (HbA1c) 7.1-11.0%
* Patients have signed the written informed consent form

Exclusion Criteria:

* Patients with type 1 diabetes mellitus (insulin¬dependent)
* Patients taking medications possibly to affect significantly the intestinal motility or the absorption of nutrients.
* Female patients who are pregnant or trying to become pregnant or lactating during the study
* Patients with alcohol, drugs or medications abuse considered by the investigator
* Patients with impaired liver function (AST, ALT>2.5× upper limit of normal)
* Patients with impaired kidney function (serum creatinine>3.0 mg/dl)
* Patients with unstable cardiovascular conditions (e.g., New York Heart Association functional class III or IV congestive heart failure or a history of myocardial infarction or stroke)
* Patients with emphysema or chronic bronchitis
* Patients with diabetic ketoacidosis
* Patients with hepatic cirrhosis
* Patients with on-going inflammatory bowel disease, colonic ulceration, partial intestinal obstruction
* Patients are predisposed to intestinal obstruction
* Patients with chronic intestinal diseases related to marked disorders of digestion or absorption
* Patients with clinically significant medical conditions that may deteriorate clinically due to gastrointestinal gas increase
* Patients with a history of lactic acidosis
* Patients with a history of allergic to repaglinide
* Patients took any hypoglycemic agent except for metformin within 3 months before study
* Patients participated investigational drug trial within 1 month before entering this study
* Patients with any other serious diseases considered by the investigator not in the condition to enter the trial

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-07

PRIMARY OUTCOMES:
change of HbA1c at 12 weeks
Change of fasting plasma glucose (FPG) at 12 weeks
Change of postprandial plasma glucose (PPG) at 12 weeks

SECONDARY OUTCOMES:
Safety parameters including adverse events such as hypoglycemia
change of liver and renal function test

CONTACTS AND LOCATIONS:
Overall Officials: T-J Wu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan